CLINICAL TRIAL: NCT06364358
Title: A Pilot to Develop and Test an Interactive Computer-adaptive Chronic Kidney Disease Education Program for Hospitalized African American Patients (I-C-CKD)
Brief Title: Interactive Computer-adaptive Chronic Kidney Disease Education Program
Acronym: ICCKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB23-0385; 5R21DK121262 (NIH)
Record Dates: First submitted 2023-05-18; First posted 2024-04-15 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases; Hypertension
Keywords: African American; Hospitalized; Patient education
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): The research assistant (RA) will use tablet to give participants baseline General Health Knowledge and Intent survey and leave printed patient education materials about general health maintenance. In the initial consent, pre-intervention survey and education materials, investigators will not provide CKD specific knowledge or inform participants about their CKD.
  Interventions: Behavioral: Usual Hospital Care
- Computerized Patient Education (Experimental): The RA will assist participants in starting the computer program and encourage review of the advanced CKD education module. The computer-adaptive education module will alter the content of education topics based on some preliminary participant information.
  Interventions: Behavioral: Computerized CKD Education

INTERVENTIONS:
Behavioral: Computerized CKD Education — The intervention is a culturally tailored computer-based adaptive program (developed during this intervention) to educate patients about kidney disease and renal replacement therapy options.
  Arms: Computerized Patient Education
Behavioral: Usual Hospital Care — Computer based patient education materials about general healthy lifestyle that will include information about the importance of a healthy diet, physical activity and medical adherence
  Arms: Usual Care

SUMMARY:
The goal of this pilot clinical trial is to evaluate a culturally tailored computerized education program in hospitalized African-American patients with advanced chronic kidney disease (CKD). The main question it aims to answer are: does computerized adaptive education (CAE) increase patients' knowledge about CKD self-care and renal replacement therapy (RRT) options compared to usual care (UC) and will CAE will be increase patients' intent to participate in CKD self-care and RRT preparation compared to UC

DETAILED DESCRIPTION:
The goal of this pilot clinical trial is to evaluate a culturally tailored adaptive computerized education program in hospitalized African-American patients with advanced chronic kidney disease (CKD). The investigator's first hypothesis is that computerized adaptive education (CAE) will be more effective than standard of care in improving knowledge about self-care for advanced CKD and renal replacement therapy (RRT) options (Primary Outcome). The primary outcome is knowledge about CKD and knowledge about RRT. The study team will measure this using the Kidney Disease Knowledge Survey (KiKs). The investigator's second hypothesis is that CAE will increase patients' intent to participate in CKD self-care (to take diabetes and/or hypertension meds, see a nephrologist, and make additional lifestyle changes like smoking cessation, exercise, low-salt diet) compared to standard of care. The study team will measure this using an investigator-developed Health Intent Survey and measure patient activation through the Patient Activation Measure (PAM). Similarly, the investigator hypothesizes that CAE will increase patients' intent to obtain non-catheter access prior to dialysis initiation, to initiate self-care dialysis (peritoneal (PD) or home hemodialysis (HHD), and/or have transplant evaluation compared to standard of care. The study team will measure this using an investigator-developed Health Intent Survey. The investigator's final hypothesis is that CAE will increase patients' action at 30 days post-discharge in participating in CKD self-care and CKD health-seeking behavior compared to standard of care controls.

ELIGIBILITY:
Inclusion Criteria:

* African-American inpatients
* Ages 18-70
* estimated glomerular filtration rate (eGFR)<45
* Enrolled in the Hospitalist Project

Exclusion Criteria:

* Does not self-identify as African American
* Not able to consent
* Unable to speak English
* eGFR <45 due to acute kidney injury
* In Intensive Care Unit
* has had a transplant
* currently on dialysis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in CKD Knowledge baseline to post patient education intervention | Baseline and 1 day post-intervention
  The Kidney Disease Knowledge Questionnaire (KIKS) is a validated instrument that assesses CKD knowledge. Scores range from 0 (no knowledge)-28 (full knowledge). Change =Post intervention-Baseline scores
Change in Knowledge about end stage kidney disease (ESKD) treatments from baseline to 1 day post patient education intervention | Baseline and 1 day post-intervention
  The Kidney Failure Treatment Knowledge is an investigator developed tool that assesses knowledge of 6 ESKD treatment options using a Likert scale (0=no knowledge and 4=a great deal of knowledge). Possible scores range from 0-24
Change in ESKD Treatment Preferences from baseline to 1 day post-intervention | Baseline and 1 day post-intervention
  The Kidney Failure Treatment Preferences Survey is an investigator developed tool that assess change in certainty of preference for each of six ESKD treatments. Scores range -12 to 12 with each question scored as -2 extremely unlikely to choose a modality to +2 extremely likely to choose a modality with a change from 0 (in any direction) as an increase in certainty.

SECONDARY OUTCOMES:
Change in Patient Activation Measure from Baseline to 30 days Post-intervention | Baseline, 1 day post-intervention, and 30 day follow-up
  The Patient Activation Measure (PAM) is a 10-item questionnaire that assesses an individual´s knowledge, skills, and confidence for managing their health and health care. The measure assesses individuals on a 0-100 scale that converts to one of four levels of activation, from low (1) to high (4). Change =Post intervention score (1 day and 30 day)-baseline score)
Increase in Health Intent baseline to post intervention (at 1 day and 30 day follow-up) | Baseline, 1 day post-intervention and 30 day follow-up
  The Health Intent Survey is an investigator-developed tool to measure participants stated intent to make healthy lifestyle changes. There are 10 questions each scored on a 5 point scale from 1=extremely unlikely to 5=extremely likely (50 total possible points with higher scores better). Change=30 day follow-up - baseline and 1 day post-intervention - baseline.
CKD Self-Management from baseline to 30 day post-intervention | Baseline and 30 day follow-up
  The CKD Self-Management Knowledge Toolkit (CKD-SMKT) is a validated 10 item survey to assess participants CKD self-management behaviors. The survey consists of 2 true /false questions for each of the 10 self-care domains and can be scored from 0 (no self-care) to 20 (full self-care). Change is 30 day score-Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Milda Saunders, MD, Principal Investigator — Associate Professor of Medicine
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Can share individual participant data (IPD) based on researcher data plan and IRB approval
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available 12 months after study completion and will remain available for 24 months
Access Criteria: Require researcher data plan and institutional review board (IRB) approval

REFERENCES:
- [Derived] King A, Omoniyi T, Zasadzinski L, Gaspard C, Gorman D, Saunders M. Interactive Computer-Adaptive Chronic Kidney Disease (I-C-CKD) Education for Hospitalized African American Patients: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Apr 17;14:e66846. doi: 10.2196/66846. PMID 40245387